CLINICAL TRIAL: NCT05224024
Title: Retzius-sparing Versus Retzius-repairing Robotic-assisted Radical Prostatectomy: A Prospective Randomized Comparison on Functional Outcomes With a 1-year Follow-up
Brief Title: Retzius-sparing Technique in Robotic-assisted Radical Prostatectomy
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Ankara University (Other)
Responsible Party: Principal Investigator, Eralp Kubilay, Medical Doctor, Ankara University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: ANKUNI641991
Record Dates: First submitted 2021-12-21; First posted 2022-02-04 (Actual); Last update posted 2022-02-04 (Actual); Status verified 2022-01

CONDITIONS: Cancer of Prostate; Prostate Adenocarcinoma; Urinary Incontinence,Stress; Erectile Dysfunction Following Radical Prostatectomy
MeSH Terms: conditions — Prostatic Neoplasms; Urinary Incontinence, Stress

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (2):
- Retzius-repairing robot-assisted radical prostatectomy group (Active Comparator): This group is randomized to operated with retzius-repairing technique as prostate cancer patients with robot assisted radical prostatectomy.
  Interventions: Procedure: Retzius-repairing robot-assisted radical prostatectomy
- Retzius-sparing robot-assisted radical prostatectomy group (Placebo Comparator): This group is randomized to operated with retzius-sparing technique as prostate cancer patients with robot assisted radical prostatectomy.
  Interventions: Procedure: Retzius-repairing robot-assisted radical prostatectomy

INTERVENTIONS:
Procedure: Retzius-repairing robot-assisted radical prostatectomy — Repairing the retzius space which is opened during the standard robot assisted radical prostatectomy.
  Other Names: Retzius-sparing robot-assisted radical prostatectomy

SUMMARY:
The objective of this study is to compare the short-term and 1-yr follow-up functional outcomes of retzius-repairing robot-assisted radical prostatectomy (RR-RARP) with retzius-sparing (RS) RARP.

This study is a single-centre, single-surgeon and a prospective randomized study.

DETAILED DESCRIPTION:
Radical prostatectomy (RP) is the standard treatment method widely used in clinically localized and locally advanced prostate cancer (PCa). The main purpose of RP is to completely remove the tumor tissue and to provide the best oncological result and as well as recovery postoperative urinary continence and erectile functions. Depending on the severity of urinary leakage, incontinence is one of the important complications that seriously affect the quality of life after RP. Robot-assisted radical prostatectomy (RARP) has become a frequently preferred surgical treatment in PCa since the early 2000s. The effort to improve functional results has led to the continuous development and evolution of the robotic technique and different approaches have been tried to achieve the best. However, no sufficient evidence was found to show the superiority of any approach. In standard RARP, there may be a risk of deterioration of anatomical structures that contribute to the urinary continence (UC) mechanism due to the need for access to the retzius space. For this purpose, in 2010, Galfano et al. described a surgical technique performed through the douglas space in RP that preserves the retzius and the structures involved in the continence mechanism. With this technique, it is aimed to provide early recovery in UC and erectile functions after surgery by protecting the retzius. In the first case series of 200 patients, it was reported that an early UC was achieved in more than 90% of the patients. In addition, it was supported by other studies that early UC recovery rates are higher with the retzius-sparing (RS) technique, and in some series, immediate UC rates at the catheter removal were reported to be higher in the RS technique. However, it was stated that there was no significant difference in 1-year results between the standard technique and the RS technique. When the current literature is reviewed, the early continence advantages of the RS technique compared to the standard technique are emphasized. On the other hand, most surgeons still have not abandoned the standard technique, and a recent questionnaire of 250 participants showed that only 11% of RARP was performed using the RS-RALP approach. Although various continence preserving techniques have been tried in the standard RARP procedure, the high quality evidence for these techniques in the literature is limited.

The focus of our study is lack of a randomized prospective study comparing the modified reconstructive anterior approach, which we define as retzius-repairing (RR), and the RS technique in the evaluation of postoperative functional outcomes. Differ from the current literature, we aim of this study is to evaluate the results of a single surgeon prospective randomized comparative study on functional outcomes at 1-year follow-up between RR-RALP and RS-RALP for clinically localized PCa treatment.

This prospective randomized study has planned to carried out between June 2021 and December 2021, after achieving the ethics committee approval. Eligible patients were randomized in a 1:1 allocation ratio and 80 consecutive patients with clinically localized PCa underwent RALP by retzius-repairing (40 patients ) and retzius-sparing (40 patients) approach by a single surgeon (KT) and surgical team at a tertiary care institution (Ankara University School of Medicine), according to a parallel design. The assignment of each patient to the first or second treatment group was randomized with a computer-based randomization table. The UC recovery rates will be evaluated at the catheter removal, and subsequently at 1, 6 and 12 months after surgery. Postoperative potency will be eveluated at 3 and 12 months after surgeries. Other outcomes are the comparisons of postoperative complication rates, positive surgical margin and 1 year oncological outcomes.

ELIGIBILITY:
Inclusion Criteria:

* Prostate cancer patients,
* Life expectancy > 10 years,
* Clinically organ confined disease (cT1-cT2),
* Biopsy Gleason score ≤ 7,
* Total serum PSA ≤ 10 ng/ml,
* Normal preoperative continence and potency.

Exclusion Criteria:

* Pre-existing urinary incontinence,
* Any previous prostatic, urethral, bladder neck surgery,
* Neoadjuvant therapy.

Sex: Male | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 80 (Estimated)
Dates: Start 2022-02-15 (Estimated); Primary Completion 2022-08-30 (Estimated); Study Completion 2022-12-31 (Estimated)

PRIMARY OUTCOMES:
Functional Outcomes-Urinary Incontinance 1st week | 1 week
  Compare two surgical technique in terms of urinary incontinence. For URINARY INCONTINANCE;
  1st week evaluation: The percentage of patients with Immediate urinary continence defined as 1 safety or no pad within 1 week of catheter removal will be compared.
Functional Outcomes-Urinary Incontinance 4th week | 4 week
  Compare two surgical technique in terms of urinary incontinence. For URINARY INCONTINANCE; 4th week evaluation will be done with International Consultation on Urinary Incontinence on Male Lower Urinary Tract Symptoms questionaire.
Functional Outcomes-Urinary Incontinance 6th month | 6 month
  Compare two surgical technique in terms of urinary incontinence. For URINARY INCONTINANCE; 6th month evaluation will be done with International Consultation on Urinary Incontinence on Male Lower Urinary Tract Symptoms questionaire.
Functional Outcomes-Urinary Incontinance 1st year | 1 year
  Compare two surgical technique in terms of urinary incontinence. For URINARY INCONTINANCE;
  1st year evaluation will be done with International Consultation on Urinary Incontinence on Male Lower Urinary Tract Symptoms questionaire.
Functional Outcomes-Erectile Dysfunction 4th week | 4 week
  For ERECTILE DYSFUNCTION; 4th week evaluation: The percentage pf patient with Immediate potency defined as erections sufficient for intercourse within the first month after surgery will be compared.
Functional Outcomes-Erectile Dysfunction 6th month | 6 month
  For ERECTILE DYSFUNCTION; 6th month evaluation will be done with International Index of Erectile Function-5 questionaire.
Functional Outcomes-Erectile Dysfunction 1st year | 1 year
  For ERECTILE DYSFUNCTION;
  1st year evaluation will be done with International Index of Erectile Function-5 questionaire.
Oncological Outcomes | 1 year
  Comparison of surgical margin positivity from pathological reports between two surgery groups.
  The percentage of partients with surgical margin positivity will be compared according to pathological investigation.

CONTACTS AND LOCATIONS:
Overall Officials: Eralp Kubilay, Principal Investigator — Ankara University
Locations (1):
- Ankara University Faculty of Medicine Urology Department, Ankara, Altındag, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Galfano A, Ascione A, Grimaldi S, Petralia G, Strada E, Bocciardi AM. A new anatomic approach for robot-assisted laparoscopic prostatectomy: a feasibility study for completely intrafascial surgery. Eur Urol. 2010 Sep;58(3):457-61. doi: 10.1016/j.eururo.2010.06.008. Epub 2010 Jun 16. PMID 20566236
- [Result] Galfano A, Di Trapani D, Sozzi F, Strada E, Petralia G, Bramerio M, Ascione A, Gambacorta M, Bocciardi AM. Beyond the learning curve of the Retzius-sparing approach for robot-assisted laparoscopic radical prostatectomy: oncologic and functional results of the first 200 patients with >/= 1 year of follow-up. Eur Urol. 2013 Dec;64(6):974-80. doi: 10.1016/j.eururo.2013.06.046. Epub 2013 Jul 8. PMID 23856036
- [Result] Galfano A, Panarello D, Secco S, Di Trapani D, Barbieri M, Napoli G, Strada E, Petralia G, Bocciardi AM. Does prostate volume have an impact on the functional and oncological results of Retzius-sparing robot-assisted radical prostatectomy? Minerva Urol Nefrol. 2018 Aug;70(4):408-413. doi: 10.23736/S0393-2249.18.03069-2. Epub 2018 Mar 28. PMID 29595042
- [Result] van der Poel HG, de Blok W, Joshi N, van Muilekom E. Preservation of lateral prostatic fascia is associated with urine continence after robotic-assisted prostatectomy. Eur Urol. 2009 Apr;55(4):892-900. doi: 10.1016/j.eururo.2009.01.021. Epub 2009 Jan 21. PMID 19171418